CLINICAL TRIAL: NCT05498662
Title: A Prospective, Observational Clinical Study of the Safety, Effectiveness and Clinical Performance of the T3 Pro Dental Implant System
Brief Title: An Observational Study of the T3 Pro Dental Implant System
Acronym: Spike
Status: Recruiting | Type: Observational
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 2201
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: T3 Pro dental implant system — treatment of tooth loss with T3 Pro dental implants

SUMMARY:
A prospective, observational, multicenter study where 60 patients needing implants in the maxilla or mandible will be enrolled. The patients will be restored with a final prosthesis no later than 4 months following implant placement surgery. The patients will come back for follow-up evaluations yearly for 2 years.

DETAILED DESCRIPTION:
This will be a prospective, observational, multicenter study. All implants will be placed in the maxilla or mandible. The patient will either have a temporary prosthesis placed (out of occlusion) immediately (during the same implant placement visit or within 48 hours) or have a temporary or definitive prosthesis placed between 3-16 weeks following implant. Final restorations for all enrolled patients will take place no later than 4 months following implant placement surgery. All restorations will utilize the full range of the ZimVie prosthetic systems. The implant system will be evaluated yearly for 2 years.

Patients who are in need of treatment with dental implants in the maxilla and/or mandible. Those patients with tooth sites having prior failed implant(s) or in need of implant revisions, or in need of major bone grafting to be done at the time of implant placement surgery are not eligible for inclusion.

A total of 60 implants, will be placed across all participating sites. It is anticipated to have 60 patients, although one patient may contribute more than 1 implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years of age
2. Patients for whom a decision has already been made to use a dental implant in an edentulous or immediately removed tooth site to be fully restored in the mandible or maxilla.
3. Site planned for immediate extraction and immediate restoration should have intact bony walls- Type I (as described in Special Procedures section) sockets as verified by CBCT and during surgery; Type II may be considered at the discretion of the treating clinician
4. Previously extracted sites (healed at least 3-4 months)
5. For all sites, presence of opposing dentition (antagonist may be natural teeth or implant supported prosthesis) that will allow for functional occlusion is essential.
6. The site intended for implant placement should have at least 10mm of alveolar bone height and sufficient restorative space for a restoration; without the need for augmentation except for minor dehiscence, which can be augmented with autogenous bone chips and/or allograft (i.e.: Puros) to improve soft tissue attachment.
7. Patients must be physically able to tolerate conventional surgical and restorative procedures (IV sedation protocols may be used at the discretion of the treating clinician).
8. Patients who provide a signed informed consent.
9. Patients who agree to be evaluated for each study visit.

Exclusion Criteria:

1. Patients with known systemic diseases such as diabetes, endocrine disease, heart disease, immuno-compromised, or mental disorders that are uncontrolled at the time of enrollment.
2. Patients with current use of bisphosphonates.
3. Patients with active infection or severe inflammation in the areas intended for treatment.
4. Patients with more than10 cigarette per day smoking habit.
5. Patients with a history of therapeutic radiation to the head or jaw.
6. Patients who are known to be pregnant at the screening visit or planning to become pregnant within 6 months of study enrollment.
7. Patients with evidence of untreated severe parafunctional habits such as bruxing or clenching.
8. Patients who have previously failed dental implants at the site intended for study implant placement
9. Patients with HIV or active Hepatitis infection.
10. Patients with a history of untreated generalized severe periodontitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Qualified patients (each patient having at least 1 tooth site treated) newly diagnosed with needing a dental implant (or more than one) in one or more tooth sites (edentulous or sick tooth in need of extraction) in the maxilla and/or mandible. Patients who have had prior implants in the treatment site that have failed (in need of revision) are not eligible for inclusion.
  *Potential study participants please note: there are costs associated with the treatment(s) provided in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Integration success/ implant survival at 2 years; primary stability | 2 years
  the lack of implant mobility observed during 2 years duration; primary stability of the implant reached during implant placement as measured by placement torque and Resonance Frequency measures

SECONDARY OUTCOMES:
Crestal bone regression | 2 years
  lack of bone loss observed and measured at 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No